CLINICAL TRIAL: NCT05677321
Title: Individual Variations of Taste and Smell Perception in Alcohol Use Disorder (AUD)
Status: Recruiting | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000421; 000421-AA
Record Dates: First submitted 2023-01-07; First posted 2023-01-10 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10-22

CONDITIONS: Alcohol Use Disorder
Keywords: chemosensation; Preference; Natural History
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with AUD: Drink regularly (i.e., 2 or more drinks per day for at least 3 days per week in the past 12 months)
- Participants without AUD: Does not drink regularly (less than 2 drinks per day for at least 3 days per week in the past 12 months)

SUMMARY:
Background:

Alcohol use disorder (AUD) is the most common substance use disorder in the world. Long-term AUD can affect a person s sense of taste and smell. This natural history study will compare alcohol drinking behaviors and measures of taste and smell in people with and without AUD.

Objective:

To understand how alcohol use changes the senses of taste and smell.

Eligibility:

People aged 18 to 65 years with or without AUD.

Design:

Participants will be screened. They will have several tests to assess their smell and taste functions. They will answer questions about their eating, alcohol use, and smoking or vaping habits.

Participants will have 2 study visits.

They will give samples of blood, nasal mucous, saliva, stool, and urine.

Their bodies will be measured. They will undergo a type of scan that uses X-rays to measure their body composition.

They will complete taste measurements. They will taste liquids by swishing them in their mouth, without swallowing. Then, they will be asked what they can detect and which flavors they preferred.

They will also complete smell measurements. They will be asked if they can identify strong odors on a metal wand. They will be asked to rate the intensity and pleasantness of odors.

Their brain activity in the frontal regions will be measured while they smell various odors. For this, we will use a brain imaging tool called functional near infrared spectroscopy.

They will have sensory testing. Sensations such as pressure, pinpricks, heat, or vibrations will be applied to their skin. Then, they will be asked what they felt.

They will keep diaries. They will write down what they eat (for 3 days), the alcohol they drink (3 days), and how much they sleep (14 days). They will wear a wristwatch-like device that records their activity for 14 days.

DETAILED DESCRIPTION:
Study Description:

This study involves comparison of taste and smell measures between individuals with and without AUD. AUD has been associated with alterations in taste and smell. These alterations are inherently concerning, regardless of whether they have any bearing on the course of other aspects of AUD. Therefore, in the proposed study we intend to assess the taste and smell differences between individuals with and without AUD. Also, we would explore the extent of taste and smell alteration in individuals with AUD and identify the biological correlates of these alterations in taste and smell.

Objectives:

AUD is a major public health concern in America. Overconsumption of alcohol is a recognized risk factor for the development of future alcohol problems. Public health efforts to modify drinking behaviors have had limited success. Not only does alcohol overuse contribute to AUD, albeit it can lead to changes in gut microbiota, as well as salivary and metabolic hormones that likely result in inflammation. Taste and smell perceptions, which can influence alcohol consumption, may differ between individuals with AUD and those without. Currently, little is known about the biomarkers related to variations in taste and smell systems in individuals with AUD. We plan to perform a series of analysis designed to investigate how individuals' variations in taste and smell perception affect alcohol consumption. We will conduct deep phenotype for taste and smell and collect blood, saliva, and nasal samples to assess the biomarkers.

Findings from this study can be used to provide evidence for future mechanistic studies to identify targets and strategies for countermeasures in preventing or improving AUD and its comorbidities. Moreover, outcomes will foster new lines of investigation for reducing risk of alcohol-related concurrent taste and smell alterations. The proposed research is aligned with the overall mission of the National Institutes of Health to promote health and disease prevention. Lastly, approaches included in this study are innovative and highly applicable to other complex health phenomena in which biological variations in inflammation and taste and smell perception impact an individual's health. This is a hypothesis-generating protocol which plays an important role at the initial stages of clinical research. We expect that the findings of the present proposed study would add some clarification to the existing contradictory reports on the chemosensory changes associated with AUD. Most importantly, this protocol is likely to help identify the differential impact of alcohol consumption on chemosensation in individuals with and without AUD.

Endpoints:

Primary Endpoint: The primary dependent measures for this study are taste and olfaction measures.

Secondary Endpoints: Secondary measures include inflammatory markers, genotypes, microbiota, salivary and metabolic hormones, biological measures, and personal factors.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

* Individuals between 18 to 65 years of age. Although the age range of participants recruited in the NIAAA Natural History protocol is between 18-77 years, due to documented knowledge that taste and smell diminishes with age, we will limit age to this range.
* Individuals with a diagnosis of AUD (for the AUD cohort) OR without a diagnosis of AUD (for the non-AUD cohort) per clinician assessment
* Able to provide their own consent.
* Due to the extensive questionnaires (administered in English language only) that participants must complete independently, fluency in the English language is needed. Hence, participants must be able to read and understand English.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Diagnosis by a medical professional of morbid obesity or BMI > 40 or renal disease.
* Any history of chronic rhinitis, eating disorder, chronic upper respiratory infection, chronic allergic rhinitis, or nasal polyps in the last 6 months of screening, or current daily use of nasal sprays.
* Altered cranial nerves associated with taste and olfaction identified by neurological evaluation during physical exam (screening visit).
* Positive pregnancy test, currently pregnant or breastfeeding.
* Hypoglycemic drug intake.
* Currently using medications known to inhibit taste response (GLP1 agonists).
* Currently experiencing temporary change/loss of taste and/or smell (individual may be rescreened when symptoms resolve).
* Persistent loss of taste and/or smell due to COVID-19 or other reason.
* NIAAA employees/staff or subordinates/relatives/co-workers of NIAAA employees/staff or study investigators.

fMRI Exclusion Criteria

* claustrophobia
* Ferromagnetic metal in the cranial cavity or eye, e.g., aneurysm clip implanted neural stimulator, cochlear implant, ocular foreign body.
* Presence of implanted cardiac pacemaker or auto-defibrillator.
* Individuals with an insulin pump.
* Presence of an irremovable body piercing.
* Individuals who are pregnant or breastfeeding during screening, or who become pregnant during the study, will be excluded from participation due to risk of exposing the fetus to undue magnetic field hazards associated with MRI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Washington D.C. area.
Sampling Method: Non-Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Taste and smell measures, alcohol drinking behavior | At enrollment
  Compare individuals with AUD to those without AUD in measures of taste and smell and alcohol drinking behaviors.

SECONDARY OUTCOMES:
Inflammatory markers, genotypes, microbiota, salivary and metabolic hormones, biological measures, and personal factors | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Paule V Joseph, C.R.N.P., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000421-AA.html